CLINICAL TRIAL: NCT03182348
Title: Coronary Optical Coherence Tomography Correlation and Strain Mapping to Investigate Human Atherosclerosis: a Feasibility Study
Brief Title: Does OCT Imaging Allow us to See Blood Vessel Development in and Around Deposits of Fat and Calcium Inside Blood Vessels
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0255
Record Dates: First submitted 2013-02-06; First posted 2017-06-09 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2020-07

CONDITIONS: Cardiovascular Disease
Keywords: Microvessels; Cardiovascular disease; OCT
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Optical coherence tomography: As part of the clinical angioplasty procedure the patient will have a coronary guidewire passed down the artery usually from the groin to the heart which is used to position balloons and stents. OCT passes over the wire in the same way. From the patients perspective the procedure may take a small amount of additional time - maximum 10-15 minutes. We would like to be able to pass a second wire down the same coronary artery called a 'buddy wire' which is sometimes required in coronary procedures. This would be used to inflate a balloon at low pressure near the area of interest in the heart in order either to exclude blood or to oppose the OCT catheter to the vessel wall if required.
  Interventions: Procedure: Optical coherence tomography

INTERVENTIONS:
Procedure: Optical coherence tomography — As part of the clinical angioplasty procedure the patient will have a coronary guidewire passed down the artery usually from the groin to the heart which is used to position balloons and stents. OCT passes over the wire in the same way. From the patients perspective the procedure may take a small amount of additional time - maximum 10-15 minutes. We would like to be able to pass a second wire down the same coronary artery called a 'buddy wire' which is sometimes required in coronary procedures. This would be used to inflate a balloon at low pressure near the area of interest in the heart in order either to exclude blood or to oppose the OCT catheter to the vessel wall if required.
  Other Names: OCT

SUMMARY:
Cardiovascular disease is the leading cause of illness and death in the world. The disease involves narrowing of blood vessels due to deposits of fat which can become coated in calcium. It is treated by percutaneous coronary intervention in which a balloon is passed down the blood vessel to remove the obstruction and where appropriate a stent is placed in the blood vessel to scaffold it.

Early stage research suggests that the growth of small blood vessels in and around the deposits of fat and calcium leads to the growth of the deposit and may contribute to plaque rupture into the vessel leading to clot formation the process which leads to heart attacks. Drugs which prevent the development of these small blood vessel restrict the development of the deposit, and those that encourage the development of these small blood vessel also increase the development of the deposit. Researchers would like to find out more about the system of blood vessels around deposits of fat and calcium in the larger blood vessels. This involves looking just beneath the surface of the blood vessel wall, and requires a detailed and accurate image. Researchers on this project would like to find out if optical coherence tomography (OCT) is a suitable technique for imaging in this way.

OCT works like an ultrasound, but using light instead of sound waves. The additional imaging will prolong the clinical procedure by 10-15 minutes.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of illness and death in the world. Central to the process of this disease is the narrowing of blood vessels due to deposits of fatty residue which can become coated in calcium. Significant narrowing of the blood vessels is treated by percutaneous coronary intervention in which a balloon is inflated and passed down the blood vessel to remove the obstruction and where appropriate a stent is placed in the blood vessel to scaffold it.

Potential participants are those who have been scheduled for a percutaneous coronary intervention, are stable, and have a diagnosis of angina pectoris, unstable angina or acute coronary syndrome. These patients will be identified and screened by their healthcare team. Potential participants will be given study information by their healthcare team, or identified to the research team who will provide study information. The initial approach may be in clinic, in hospital, or by post.

Participants will be asked to give written informed consent to participate in the study. At the clinical pre-procedure visit consent is sought, exclusion and inclusion criteria checked.

Procedure: On the day of the patients procedure they will receive standard clinical care comprising angiography (imaging of the blood vessel), angioplasty (removal of fatty deposits with a balloon) and stenting. Before and after the procedure the patient will receive medication and after care as per standard clinical care. Those patients who are clinically indicated for stenting will undergo OCT imaging prior to the angioplasty and stenting.

The researchers need to allow flexibility in the process of acquiring the OCT images, so they can optimize the quality of the image. Therefore, the speed of pullback (removal of the catheter) and choice of blood clearing agents will not be pre-specified. Serial images of the same part of the vessel may be taken.

As part of the clinical angioplasty procedure the patient will have a coronary guidewire passed down the artery usually from the groin to the heart which is used to position balloons and stents. OCT passes over the wire in the same way. From the patients perspective the procedure may take a small amount of additional time - maximum 10-15 minutes. We would like to be able to pass a second wire down the same coronary artery called a 'buddy wire' which is sometimes required in coronary procedures. This would be used to inflate a balloon at low pressure near the area of interest in the heart in order either to exclude blood or to oppose the OCT catheter to the vessel wall if required.

If a patient returns for subsequent percutaneous coronary intervention they will be invited to participate again.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective percutaneous coronary intervention or coronary angiography with a view to coronary intervention on routine clinical criteria with diagnosis of angina pectoris, unstable angina or acute coronary syndrome with angiographically significant stenosis(es) (>70%) of one or more native coronary arteries.

Exclusion Criteria:

* Primary angioplasty for S T -elevation myocardial infarction. Clinically unstable patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective percutaneous coronary intervention or coronary angiography with a view to coronary intervention on routine clinical criteria with diagnosis of angina pectoris, unstable angina or acute coronary syndrome with angiographically significant stenosis(es) (>70%) of one or more native coronary arteries.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Markers of high risk coronary diseases | through study completion, an average of 1 year (Aprox March 2018)
  Novel OCT features as potential markers of high risk coronary diseases

CONTACTS AND LOCATIONS:
Overall Officials: David Adlam, BA,BM,BCH,DPhil,MRCP, Principal Investigator — NIHR Leicester Cardiovascular BRU
Locations (1):
- NIHR Cardiovascular BRU, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No